CLINICAL TRIAL: NCT07188857
Title: Study on the Relationship Between Opioid Drugs and the Therapeutic Efficacy of Immunotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Hubei Cancer Hospital (Other)
Collaborators: Cancer Hospital Chinese Academy of Medical Science (Unknown)
Responsible Party: Principal Investigator, Yu Qian, Doctor, Hubei Cancer Hospital
Other Study IDs: OPIOIDS
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Pain Management; Immune Checkpoint Inhibitor; Opioid
Keywords: pain management; opioids; immune checkpoint inhibitor
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- immunotherapy group with opioids: immunotherapy group with opioids
- immunotherapy group without opioids: immunotherapy group without opioids

SUMMARY:
Relationship between pain and the efficacy of immunotherapy: Does the degree of pain control affect the therapeutic efficacy of ICIs? Does the use of opioid drugs independently affect the efficacy of immunotherapy?

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years; Histologically confirmed advanced NSCLC (Stage IIIb-IV); Need to receive ICIs treatment; Accompanied by moderate or severe pain (NRS score ≥ 4); Need to use opioid drugs for pain management; Able to understand and sign the informed consent form.

Exclusion Criteria:

* Suffering from severe dysfunction of important organs such as heart, liver, and kidney; Suffering from mental illness or receiving treatment with psychotropic drugs; Pregnant or lactating women; Participating in other clinical trials; Allergic to opioid drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital based study
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-17 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
The relationship between different degrees of pain control and the therapeutic efficacy of ICIs (immune checkpoint inhibitors) in patients with advanced cancer pain. | From enrollment to the end of treatment at 8 weeks
  The therapeutic efficacy includes progression-free survival (PFS), objective response rate (ORR), and overall survival (OS). Additionally, analyze whether the use of opioid drugs independently affects the therapeutic efficacy.

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years after the publication of results